CLINICAL TRIAL: NCT05332730
Title: A Randomized, Double-blind, Single-dose, Parallel Three-arm Comparative Study on Pharmacokinetics and Safety of BAT2506 Injection Versus the EU-licensed and US-licensed Simponi® in Healthy Chinese Male Subjects
Brief Title: A Study on Pharmacokinetics and Safety of BAT2506 Injection Versus Simponi®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2506-003-CR
Record Dates: First submitted 2022-03-03; First posted 2022-04-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT2506 (Experimental): BAT2506 injection, 50 mg, subcutaneous administration. Dose regimen: 50 mg/0.5 mL/syringe, subcutaneously injected at the lower abdomen, except for the 5 cm area around the navel. Do not inject into skin that is tender, bruised, red, scaly, or hard. Avoid areas with scars or stretch mark.
  Interventions: Drug: BAT2506 injection
- Simponi® (EU commercially available product) (Active Comparator): 50 mg, subcutaneous administration Dose regimen: 50 mg/0.5 mL/syringe, subcutaneously injected at the lower abdomen, except for the 5 cm area around the navel. Do not inject into skin that is tender, bruised, red, scaly, or hard. Avoid areas with scars or stretch mark.
  Interventions: Drug: Simponi® (EU commercially available product)
- Simponi® (US commercially available product) (Active Comparator): 50 mg, subcutaneous administration Dose regimen: 50 mg/0.5 mL/syringe, subcutaneously injected at the lower abdomen, except for the 5 cm area around the navel. Do not inject into skin that is tender, bruised, red, scaly, or hard. Avoid areas with scars or stretch mark.
  Interventions: Drug: Simponi® (US commercially available product)

INTERVENTIONS:
Drug: BAT2506 injection — 50 mg, subcutaneous administration
  Arms: BAT2506
Drug: Simponi® (EU commercially available product) — 50 mg, subcutaneous administration
  Arms: Simponi® (EU commercially available product)
Drug: Simponi® (US commercially available product) — 50 mg, subcutaneous administration
  Arms: Simponi® (US commercially available product)

SUMMARY:
This is a randomized, double-blind, parallel three-arm, and single-dose Phase I clinical study, designed to compare the similarity of pharmacokinetics, safety and immunogenicity between BAT2506 Injection and Simponi® (EU-licensed and US-licensed) after single subcutaneous administration in healthy Chinese male subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel three-arm, and single-dose Phase I clinical study, designed to compare the similarity of pharmacokinetics, safety and immunogenicity between BAT2506 Injection and Simponi® (EU-licensed and US-licensed) after single subcutaneous administration in healthy Chinese male subjects.

The study planes to enroll 375 healthy male subjects who will be randomly assigned to the BAT2506 Injection group, Simponi® (EU-licensed) or Simponi® (US-licensed) groups in a 1:1:1 ratio to receive a single subcutaneous injection of 50 mg BAT2506 Injection or Simponi® (EU-licensed or US-licensed).

ELIGIBILITY:
Inclusion Criteria:

* 1)Signed the ICF and fully understood the trial conduction, procedure and potential adverse reactions before included the trial;
* 2)Able to complete the study in accordance with the requirements of the protocol;
* 3)Subjects (including their partners) who are willing to refrain from pregnancy and will not donate sperm throughout the trial and within 6 months after the end of the study, and willing to take effective contraceptive method, see Appendix 4 for specific contraceptive methods;
* 4)Healthy male subjects at age of 18-55 years with a body mass index (BMI) between 18 and 28 kg/m2 (inclusive) and a body weight between 50 and 80 kg (inclusive);
* 5)Subjects with normal physical examination and vital signs or non-clinically significant abnormalities.

Subjects with normal abdominal color Doppler ultrasound, laboratory tests and other examination results or non-clinically significant abnormalities.

Exclusion Criteria:

* 1)Subjects who smoked more than 5 cigarettes every day within 3 months prior to the trial;
* 2)Subjects with a history of allergies to the study drug, or subjects with allergic constitution (allergic to a variety of drugs and foods);
* 3)Subjects with a history of alcohol abuse (consuming 14 or more units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
* 4)Subjects who donated blood within 3 months prior to screening or plan to donate blood during the study period;
* 5)Subjects who had major injuries or underwent surgery or had fractures within 4 weeks prior to enrollment, or who are scheduled to undergo surgery during the study period;
* 6)Subjects whose abnormalities in past medical history are clinically significant or other clinical findings suggest the following clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, blood, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular diseases);
* 7)Subjects who suffered from malignant tumors (excluding those with basal cell carcinoma which has been surgically resected);
* 8)Subjects with clinically significant chronic or acute infections at screening/enrollment, or with active infections, including acute and chronic infections and local infections (bacteria, viruses, parasites, fungi or other pathogens of opportunistic infectious diseases);
* 9)Patients having a history of tuberculosis, or having latent tuberculosis infection or clinically suspected tuberculosis (including but not limited to pulmonary tuberculosis);
* 10)Subjects who have contacted with tuberculosis patients or/and had symptoms and/or signs suspected of being tuberculosis within 3 months prior to screening ;
* 11)Subjects who have used Simponi®, any anti-tumor necrosis factor (TNF-α) biologic, or have used any biologics or monoclonal antibodies within 6 months prior to enrollment ;
* 12)Subjects who have used drugs (including but not limited to prescription drugs, traditional Chinese medicines, over-the-counter drugs, etc.) within 30 days prior to enrollment ;
* 13)Subjects who have participated in other drug clinical trials within 3 months prior to enrollment;
* 14)Have received live vaccine within 12 weeks prior to study administration or plan to receive live vaccine during study period; Have received inactivated vaccine (including COVID-2019 inactivated vaccine) within 2 weeks prior to administration or plan to receive inactivated vaccine during study period.
* 15)Subjects with a history of hypertension or systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg at screening/enrollment, which is judged to be a clinically significant abnormality;
* 16)Subjects with clinically significant abnormalities in ECG;
* 17)Positive hepatitis B surface antigen at screening [or negative hepatitis B surface antigen and meeting all three of the following: positive hepatitis B core antibody, negative hepatitis B surface antibody, and hepatitis B virus deoxyribonucleic acid (HBV DNA) levels exceed the normal quantification range]; or positive hepatitis C antibody, hepatitis C core antigen, HIV antigen/antibody, or positive syphilis spirochete antibody;
* 18)Subjects with clinically significant abnormalities in frontal chest radiography;
* 19)Those who have tested positive for enzyme-linked immunospot assay (T-SPOT. TB);
* 20)Subjects who have taken any alcoholic products within 24 hours prior to the use of the study drugs;
* 21)Those who have tested positive for drug abuse or have a history of drug abuse within past five years;
* 22)Ineligible subjects based on investigator's judgment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — (1) healthy subjects are free from underlying diseases and concomitant medications, so that the PK parameters of all individuals tend to be more consistent; (2) the inclusion of male subjects can exclude the influence of female menstrual cycle, thereby reducing the interference from the fluctuations of PK parameters among subjects. Under the premise of fully considering the safety of the subjects, this study chooses healthy male subjects as the test population.
Enrollment: 375 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Cmax | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Peak plasma concentration
AUC0-∞ | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  area under the drug concentration-time curve

SECONDARY OUTCOMES:
(AUC0-t) | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Area under the drug concentration-time curve from time 0 to the last quantifiable data point
temperature | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal temperature findings
pulse | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal pulse findings
blood pressure | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal blood pressure findings
skin mucosa | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal skin mucosa findings
lymph nodes | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal lymph nodes findings
head and neck | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal head and neck findings
chest | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal chest findings
abdomen | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal abdomen findings
spine/extremities | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal spine/extremities findings
heart rate | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal heart rate findings
PR Interval | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal PR Interval findings
RR Interval | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal RR Interval findings
QRS Interval | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal QRS Interval findings
QT Interval | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal QT Interval findings
QTc interval | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  number of participants with abnormal QTc Interval findings
hematology, | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Number of participants with abnormal hematology findings
biochemistry | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Number of participants with abnormal biochemistry findings
coagulation routine | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Number of participants with abnormal coagulation routine findings
urinalysis | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Number of participants with abnormal urinalysis findings
Injection-site reaction Injection-site reaction | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Injection-site reaction Adverse events (AE), serious adverse events (SAE), etc.
Adverse events (AE) | on Day1,2,3,4,5,6, 7, 8, 9, 15, 22, 29, 36, 43, 50, 57, 64, and 78
  Adverse events (AE), serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jinlin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No